CLINICAL TRIAL: NCT01960296
Title: Evaluation of Clopidogrel Use in Peri-Operative General Surgery Patients: A Prospective Study
Brief Title: Does Continued Use of Clopidogrel Into Surgery Cause Increased Perioperative Bleeding?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 10-1067
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Clopidogrel
Keywords: clopidogrel; general surgery
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): Continue home dose of clopidogrel into surgery
  Interventions: Drug: Clopidogrel
- Discontinue (Active Comparator): Discontinue home dose of clopidogrel one week before surgery. Resume after surgery.
  Interventions: Drug: Discontinue Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Continue home dose of clopidogrel into surgery
  Arms: Clopidogrel
Drug: Discontinue Clopidogrel — Discontinue home dose of clopidogrel one week before surgery. Resume after surgery.
  Arms: Discontinue

SUMMARY:
Patients who on taking clopidogrel are randomized to either continue clopidogrel into general surgery or discontinue clopidogrel 7 days before surgery. All patients resume clopidogrel after surgery. The investigators track the development of bleeding complications that may develop within 90 days of the surgery. Patients are medically cleared to be in either arm of the study by their cardiologist and surgeon. There is currently no evidence to support for or against the use continuation or discontinuation of clopidogrel prior to general surgery.

DETAILED DESCRIPTION:
A medical record review was performed of 104 consecutive patients undergoing general surgical procedures while receiving antiplatelet therapy. Patients were identified from an administrative database by crossreferencing clopidogrel with abdominal operative procedures. The records of only patients who were actively receiving antiplatelet therapy, with the last clopidogrel dose within 45 days of their operation, were considered in the study.

ELIGIBILITY:
Inclusion Criteria:

* taking clopidogrel
* undergoing general surgery
* cleared by both cardiologist and surgery for randomized arm

Exclusion Criteria:

* previous history of bleeding complications/bleeding disposition
* no capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celia M Divino, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Chernoguz A, Telem DA, Chu E, Ozao-Choy J, Tammaro Y, Divino CM. Cessation of clopidogrel before major abdominal procedures. Arch Surg. 2011 Mar;146(3):334-9. doi: 10.1001/archsurg.2011.23. PMID 21422366
- [Result] Chu EW, Chernoguz A, Divino CM. The evaluation of clopidogrel use in perioperative general surgery patients: a prospective randomized controlled trial. Am J Surg. 2016 Jun;211(6):1019-25. doi: 10.1016/j.amjsurg.2015.05.036. Epub 2015 Aug 20. PMID 27002953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from 6 institution-affiliated ambulatory general surgery clinics were assessed for eligibility between January 2011 and May 2013.
Period: Overall Study
Arm/Group | Clopidogrel | Discontinue
Started | 23 | 25
Completed | 21 | 22
Not Completed | 2 | 3
Not completed — Postponed surgery | 1 | 0
Not completed — Received different procedure | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel | Discontinue | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (0) | 67.9 (0) | 67.9 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 14 | 13 | 27
Indication [Number; unit: participants]
  Coronary stent | 18 | 13 | 31
  CVA | 1 | 2 | 3
  Other | 2 | 7 | 9
CAD/CVD/PAD [Number; unit: participants] — Coronary Artery Disease(CAD)/Cerebrovascular Disease(CVD)/Peripheral Arterial Disease(PAD)
  participants
    yes | 20 | 18 | 38
    no | 1 | 4 | 5
Hypertension [Number; unit: participants]
  yes | 19 | 19 | 38
  no | 2 | 3 | 5
Diabetes [Number; unit: participants]
  yes | 12 | 12 | 24
  no | 9 | 10 | 19
HL [Number; unit: participants]
  yes | 19 | 20 | 39
  no | 2 | 2 | 4
ASA score [Number; unit: participants] — Preoperative American Society of Anesthesia (ASA) scores to evaluate the degree of a patient's "sickness" or "physical state" before selecting the anesthetic or before performing surgery, with one being normal to five being severely impaired.
  participants
    2 | 4 | 1 | 5
    >2 | 17 | 21 | 38
Normal platelet function [Number; unit: participants]
  yes | 15 | 16 | 31
  no | 6 | 6 | 12
Aspirin Use [Number; unit: participants]
  yes | 14 | 18 | 32
  no | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Bleeding-related Re-hospitalization
Description: Perioperative Bleeding Complications as indicated by bleeding requiring re-admission.
Time Frame: up to 90 days post op
Measure: Number; unit: participants
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 21 | 22
participants | 1 | 1

2. Secondary Outcome: Procedure Estimated Blood Loss
Time Frame: up to 90 days postop
Population: Quantitative estimation of blood loss was available in 31 of the 43
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 14 | 17
mL | 73.6 (24.9) | 52.1 (18.8)

3. Primary Outcome: Perioperative Bleeding Complications
Description: Development of perioperative bleeding complications as indicated for need for blood transfusions, hematoma, and bleeding requiring re-operation.
Time Frame: up to 90 days postop
Measure: Number; unit: participants
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 21 | 22
participants | 0 | 0

4. Secondary Outcome: Procedure Time
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 21 | 22
minutes | 114.3 (11.3) | 100.4 (12.7)

5. Secondary Outcome: Average Change in Hematocrit
Description: hematocrit levels change from preoperative to postoperative
Time Frame: baseline and Day 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 21 | 22
percent change | -3 (0.6) | -1 (0.8)

6. Secondary Outcome: Average Length of Hospital Stay
Time Frame: up to 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 21 | 22
days | 2.2 (0.6) | 2.4 (1.1)

7. Secondary Outcome: Same Day Discharged
Description: Number of patients discharged on the day of surgery
Time Frame: up to 90 days
Measure: Number; unit: participants
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 21 | 22
participants
  same day discharged | 8 | 12
  hospital admission | 13 | 10

8. Secondary Outcome: Development of Myocardial Infarction or Thrombosis
Time Frame: up to 90 days
Measure: Number; unit: participants
Arm/Group | Clopidogrel | Discontinue
Number analyzed (Participants) | 21 | 22
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Clopidogrel | Discontinue
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=21) | Discontinue (N=22)
Intra-abdominal hematoma (Surgical and medical procedures) | 1 (1) | 1 (1) — Readmission for percutanenous drainage without requiring re-operation

LIMITATIONS AND CAVEATS:
The major limitation of the study is its low sample size, making it underpowered to draw unequivocal conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes